CLINICAL TRIAL: NCT06670443
Title: Electrical Stimulation for Respiratory and Leg Muscles Impact on Pulmonary Function and Leg Restless Syndrome in COPD Patients
Brief Title: Electrical Stimulation for Respiratory and Leg Muscles Impact on COPD Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, marwa mahmoud elsayed mahmoud, Assistant Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/005638
Record Dates: First submitted 2024-10-31; First posted 2024-11-01 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Intervention group: active NMES (350 μs pulses - 50 Hz frequency) will be applied at the lower third of the thigh, just above the patella, and the proximal electrode 5-10 cm below the anterior superior iliac spine for quadriceps muscle stimulation, and for intercostal muscles stimulation, NMES will be bilateral, parallel to the ribs, in the intercostal space. The proximal electrode will be positioned close to the sternum, and the distal electrode laterally, close to the midaxillary line. In addition to conventional pulmonary rehabilitation program that comprised diaphragmatic and pursed lips breathing
  Interventions: Device: experimental group
- control group (Placebo Comparator): control group: placebo NMES at the same points in addition to the same conventional pulmonary rehabilitation program
  Interventions: Device: control group

INTERVENTIONS:
Device: experimental group — Electrical neuromuscular stimulation electrode patches will be applied over the intercostal respiratory muscles and leg muscles (placed superficially just below each knee, over the head of the fibula, in close proximity to the common peroneal nerve).
  Other Names: NMES
  Arms: experimental group
Device: control group — Placebo electrical neuromuscular stimulation electrode patches will be applied over the intercostal respiratory muscles and leg muscles (placed superficially just below each knee, over the head of the fibula, in close proximity to the common peroneal nerve).
  Other Names: placebo NMES
  Arms: control group

SUMMARY:
Electrical neuromuscular stimulation electrode patches will be applied over the intercostal respiratory muscles and leg muscles In addition to conventional pulmonary rehabilitation

DETAILED DESCRIPTION:
Intervention group: active NMES (350 μs pulses - 50 Hz frequency) will be applied at the lower third of the thigh, just above the patella, and the proximal electrode 5-10 cm below the anterior superior iliac spine for quadriceps muscle stimulation, and for intercostal muscles stimulation, NMES will be bilaterally, parallel to the ribs, in the intercostal space. The proximal electrode will be positioned close to the sternum, and the distal electrode laterally, close to the midaxillary line. In addition to conventional pulmonary rehabilitation program that comprised diaphragmatic and pursed lips breathing.

control group: placebo NMES at the same points in addition to the same conventional pulmonary rehabilitation program

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoes four main clinical criteria for the diagnosis of RLS according to the international restless leg syndrome study group (IRLSSG) including

  1. an urge to move legs that is usually associated with paresthesia.
  2. alleviation of the symptoms by moving the legs.
  3. aggravation or exacerbation of the symptoms particularly at rest or during sitting or lying down in the bed.
  4. worsening of the signs at night. patients with diagnosed with grade I and grade II COPD their ages ranged between 45-55 o All patients will be clinically and medically stable when attending the study

Exclusion Criteria:

* History of Deep venous thrombosis

  * History of Bleeding disorders
  * Have an implantable device like a pacemaker
  * Recent Infected wound
  * History of allergic response to the electrodes, gel or tape
  * patients who participating in any other exercise program
  * Loss of sensation or numbness

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-10 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
dynamic gait index | 10 weeks
  It will be measured by dynamic gait index which includes eight items, walking on level surfaces, changing speeds, head turns in horizontal and vertical directions, walking and turning 180 degrees to stop, stepping over and around obstacles, and stair ascent and descent. Each item is scored on a scale of 0 to 3, with 3 indicating normal performance and 0 representing severe impairment. The best possible score on the DGI is a 24

SECONDARY OUTCOMES:
pulmonary functions | 10 weeks
  It will be measured by spirometry to assess forced expiratory volume in the first second (FEV1), forced vital capacity (FVC), and FEV1/FVC. The patient is instructed to take in a deep breath and then, as fast as he can, blow out all the air into a tube connected to a machine (spirometer). To get the "best" test result, the test is repeated three times.
Dyspnea | 10 weeks
  It will be assessed by modified Borg dyspnea scale which uses a scale from 0 to 10, where 0 represents no dyspnea and 10 represents maximal dyspnea
International restless leg syndrome questionnaire | 10 weeks
  Developed as a tool for assessing the severity Restless Legs Syndrome (RLS), the 10-item questionnaire asks respondents to use Likert-type ratings to indicate how acutely the disorder has affected them over the course of the past week. Questions can be divided into one of two categories: disorder symptoms (nature, intensity, and frequency) and their impact (sleep issues, disturbances in daily functioning, and resultant changes in mood) Rating scale and the RLS will be evaluated using the lower-limit clinical definition issued by the IRLSSG. Respondents with four "yes" were treated as having RLS. Respondents further performed the IRSSG Severity Scale with ten items to determine the severity of RLS symptoms. Patients were categorized into four classes of RLS ratings: mild (0~10), moderate (11~20), extreme (21~30), and very serious (31~40)
visual analogue scale | 10 weeks
  the pain will be evaluated by visual analogue scale (VAS) which assess pain intensity and progression. It is a straight horizontal line of fixed length, usually 100 mm. The ends are defined as the extreme limits of the parameter to be measured (symptom, pain, health) orientated from the left (worst) to the right (best).
Sleep quality | 10 weeks
  It will be examined by pittsburgh sleep quality index (PSQI) which is a self-report questionnaire that assesses sleep quality over a 1-month time interval. It consisted of 19 items, the PSQI measures several different aspects of sleep, offering seven component scores and one composite score. The component scores consist of subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction.
  Each item is weighted on a 0-3 interval scale. The global PSQI score is then calculated by totaling the seven component scores, providing an overall score ranging from 0 to 21, where lower scores denote a healthier sleep quality
Chronic Respiratory Disease Questionnaire | 10 weeks
  Qol will be evaluated by The Chronic Respiratory Disease Questionnaire (CRQ) is a disease-specific health-related quality of life questionnaire. It was developed to measure the impact of Chronic Obstructive Pulmonary Disease (COPD) on a person's life. It consists of 20 items across four dimensions: dyspnea, fatigue, emotional function, and mastery. Items in each section are scored from 1 (most severe) to 7 (no impairment).

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy, Dokki, Egypt